CLINICAL TRIAL: NCT06326749
Title: Investigation of the Effect of Modified Graded Motor Imagery Training on Upper Extremity Motor Function, Activities of Daily Living, Quality of Life and Motor Imagery Skills in Stroke Patients
Brief Title: Effectiveness of Modified Graded Motor Imagery Training in Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Havva Adlı, lecturer, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/19
Record Dates: First submitted 2024-03-10; First posted 2024-03-22 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Graded Motor Imagery; Stroke; Action Observation Training; Motor Imagery
Keywords: graded motor imagery; action observation training; Stroke; hemiplegia; upper limb function; activities of daily living; life quality
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Modified Graded Motor Imagery and Conventional Treatment Group: (Experimental): The modified DMI program consists of 4 stages: lateralization, open motor imagery including action observation training, mirror therapy and upper extremity functional exercise. The program will be implemented for 8 weeks, 3 days a week, under the supervision of a physiotherapist. Lateralization training will be applied in the first 2 weeks. Motor imagery training will be implemented in the 3rd and 4th weeks. For the second stage, the application will be combined with action observation training. As the 3rd stage, mirror therapy will be performed in the 5th and 6th weeks. The participant will be asked to perform some exercises while watching the reflection of the intact extremity in the mirror. In the final stage, they will be asked to physically perform upper extremity functional exercises. The total treatment time will be 40-50 minutes, with patients receiving 20-30 minutes of modified grade motor imagery and 20 minutes of conventional treatment.
  Interventions: Other: Modified Graded Motor Imagery and Conventional Treatment Group
- Graded Motor Imagery and Conventional Treatment Group: (Experimental): The DMI program consists of 3 stages: lateralization, open motor imagery and mirror therapy. The program will be implemented for 8 weeks, 3 days a week, under the supervision of a physiotherapist. First, lateralization training will be applied. In the second stage, motor imagery training will be applied. This phase will be carried out in a quiet environment by asking the participants to fully focus on the visualization of the movements. Two methods will be used for the imagined movements. In particular, visuals of the shoulder and hand used in the lateralization phase will be used to visualize movements related to the normal movement of the upper extremity. Participants will also be asked to imagine different activities in daily life. In the final stage, mirror therapy will be applied. The participant will be asked to perform some exercises while watching the reflection of the intact extremity in the mirror.
  Interventions: Other: Graded Motor Imagery and Conventional Treatment Group
- Conventional Treatment Group: (Experimental): Within the scope of the conventional treatment Bobath Method, facilitating movement and functional activities in the upper and lower extremities, activating trunk muscles, facilitating basic functional activities such as turning in bed, coming to sit and standing, improving weight bearing while sitting and standing, postural control, balance and walking. A targeted exercise program will be created. In line with this goal, upper and lower extremity exercises; don't turn around, don't come to sit, don't stand up; Exercises to activate core muscles; such as bridging, functional reaching; weight bearing and balance training; It is planned to implement walking training. Treatment time will be 40-50 minutes.
  Interventions: Other: Conventional Treatment Group

INTERVENTIONS:
Other: Modified Graded Motor Imagery and Conventional Treatment Group — A modified form of graded motor imagery training and conventional rehabilitation will be applied.
  Arms: Modified Graded Motor Imagery and Conventional Treatment Group:
Other: Graded Motor Imagery and Conventional Treatment Group — Graded motor imagery training and conventional rehabilitation will be applied.
  Arms: Graded Motor Imagery and Conventional Treatment Group:
Other: Conventional Treatment Group — conventional rehabilitation will be applied.
  Arms: Conventional Treatment Group:

SUMMARY:
In the study, movement observation training, Modified Graded Motor Imaging Training, which includes upper extremity functional exercises, and Graded Motor Imaging Training, where the standard protocol is applied, will be used in stroke patients to improve their upper extremity motor functions and daily lives. It is aimed to present it on an evidence-based basis by investigating its effects on Daily Living Activity, quality of life, upper extremity-specific right/left lateralization performance, mental stopwatch performance and motor imagery skills.

DETAILED DESCRIPTION:
At study is planned as a combination of action observation training, motor imagery and graded motor imagery training, which have come to the fore in recent years and whose importance increases with each passing year. Additionally, its preferability in treatment will be investigated by comparing it with Graded Motor Imagery training, in which the standard protocol is applied. It is anticipated that treatment protocols will shed light on future studies.

The hypotheses of the study are as follows:

Hypothesis 1: Modified Graded Motor Imagery training is more effective than Graded Motor Imagery training and conventional treatment in improving upper extremity motor functions in individuals with stroke.

Hypothesis 2: Modified Graded Motor Imagery training is more effective than Graded Motor Imagery training and conventional treatment in improving daily living activities in individuals with stroke.

Hypothesis 3: Modified Graded Motor Imagery training is more effective than Graded Motor Imagery training and conventional treatment in improving the quality of life in individuals with stroke.

Hypothesis 4: Modified Graded Motor Imagery training is more effective than Graded Motor Imagery training and conventional treatment in improving motor imagery skills in individuals with stroke. Design of the study: The study was designed as a randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

Hemiplegia was observed after CVO, According to the Edinburgh Handedness Questionnaire, those who actively use their right extremity, Those with right hemisphere involvement, Those aged 18 and over, Having been diagnosed with stroke at least 1 month ago and at most 6 months ago, Middle cerebral artery involvement, Having a Standardized Mini Mental Test score of 24 or above, having a Stage 2b or above according to Eggers staging, Able to actively control hands, wrists and fingers and perform the release reflex Those who want to participate in the study voluntarily and Individuals with informed consent will be included in the study.

Exclusion Criteria:

Those with major neurological, orthopedic or rheumatological disorders that affect upper extremity function other than stroke (Polyneuropathy, Parkinson's, Multiple Sclerosis, Rheumatoid Arthritis, etc.).

Those with upper extremity amputation, Uncontrolled arrhythmia, uncontrolled hypertension, unstable cardiac status Active malignancy and receiving chemo/radiotherapy related to it Uncooperative due to aphasia or cognitive impairment Individuals with vision and hearing problems Having a communication problem that may prevent implementation of the evaluations and/or treatment program Individuals who do not allow mental evaluation, cannot fill out the scales, and are illiterate will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity Motor Rating Scale | before treatment, 2 months, 4 months
  The scale is a widely used, reliable and valid test to evaluate paretic upper extremity motor impairment in stroke patients. From this scale, where each parameter is scored between 0-2 points, a maximum score of 66 can be obtained, and high scores indicate good motor functions.
Wolf Motor Function Test (WMFT) | before treatment, 2 months, 4 months
  WMFT is used to evaluate motor skill in patients with upper extremity motor dysfunction. The 15 functional activities evaluated are scored between 0-5 points and the functional skill score is calculated by taking the average of the total score. Higher scores indicate better functional ability. In the performance time section, how long each activity took is recorded. A maximum of 120 seconds is allowed to complete an activity. If the activity cannot be completed within this time, the performance time is recorded as 120 seconds.
Modified Barthel Index | before treatment, 2 months, 4 months
  MBI, which is used to measure the independence of individuals in daily living activities, emerged by modifying the Barthel Index. MBI includes 10 items related to activities of daily living. Total score is between 0-100. As the score increases, individuals' independence in daily living activities increases.
Stroke-Specific Quality of Life Scale | before treatment, 2 months, 4 months
  It consists of a total of 49 items for 12 subcategories (mobility, fitness, upper extremity functionality, work/productivity, mood, self-care, social roles, family roles, language, vision, thinking and personality) that evaluate the quality of life of individuals with stroke. The higher the total score, the better the stroke individual's quality of life.

SECONDARY OUTCOMES:
Lateralization Assessment | before treatment, 2 months, 4 months
  Right/left lateralization performance of the upper extremity will be evaluated with the "Recognise™" application developed by the Neuro Orthapedic Institute. The "Recognise™ Hand" and "Recognise™ Shoulder" sections of this application and the "Vanilla" part of these sections will be used. Accuracy rates and reaction time in the application will be recorded. An increase in the accuracy rate indicates that lateralization performance has improved.
Mental Chronometry Time | before treatment, 2 months, 4 months
  It will be used to evaluate the chronometric aspect of motor imagery. You will be given the task of wearing and folding a T-shirt for the mental stopwatch period.First, the motor imagery task will be performed. The time written on the screen is recorded by the observer. For the physical phase of the test, the same application is actually carried out and the time is recorded with the help of a stopwatch. Mental stopwatch rate will be calculated.
  Mental stopwatch ratio = (Time in which the movement is physically performed - Time in which the movement is performed with imagination) / Time in which the movement is physically performed.
Kinesthetic and Visual Imagery Questionnaire (KGIA) | before treatment, 2 months, 4 months
  CSIA will be used to evaluate motor imagery skills. After experiencing the movement in reality, he will be asked to imagine himself watching the same movement as if it were actually performed. Participants will evaluate the quality of the image in the visualization by giving points between 1 and 5, including "1 (no image)" and "5 (clear as the original)". An increase in the score indicates improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braun N, Kranczioch C, Liepert J, Dettmers C, Zich C, Busching I, Debener S. Motor Imagery Impairment in Postacute Stroke Patients. Neural Plast. 2017;2017:4653256. doi: 10.1155/2017/4653256. Epub 2017 Mar 28. PMID 28458926
- [Background] Candiri B, Talu B, Guner E, Ozen M. The effect of graded motor imagery training on pain, functional performance, motor imagery skills, and kinesiophobia after total knee arthroplasty: randomized controlled trial. Korean J Pain. 2023 Jul 1;36(3):369-381. doi: 10.3344/kjp.23020. Epub 2023 Jun 22. PMID 37344366
- [Background] Yu JA, Park J. The effect of first-person perspective action observation training on upper extremity function and activity of daily living of chronic stroke patients. Brain Behav. 2022 May;12(5):e2565. doi: 10.1002/brb3.2565. Epub 2022 Apr 10. PMID 35398981